CLINICAL TRIAL: NCT06089720
Title: An Antimicrobial Effect of ZnO Nanoparticles Coated Orthodontic Molar Tube (A Randomized Clinical Trial)
Brief Title: ZnO Nanoparticles Coated Orthodontic Molar Tube
Acronym: ZnONPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Kamil Jawad, Doctor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 782423
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Evaluations, Diagnostic Self; Antimicrobial; Orthodontic Appliance Complication; Bacterial Overgrowth; Dental White Spot; Plaque Induced Gingivitis; Plaque, Dental
Keywords: Nanoparticles; zinc oxide nanoparticle; coating; orthodontic molar tube; electrophoretic deposition cell; EPD CELL; nanomaterials; antimicrobial effect; bacterial culture
MeSH Terms: conditions — Dental Caries; Dental Plaque

STUDY DESIGN:
Intervention Model Description: 72 orthodontic molar tubes will be divided in two groups control 36 uncoated OMT, and 36 experimental groups that will receiving the zinc oxide nanoparticle coating.
Who Masked: Participant, Outcomes Assessor
Masking Description: When applications of orthodontic molar tubes to patients mouth through routine orthodontic treatment, the clinicians will explain the procedure to patients without knowing the about which side coated or not .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc oxide nanoparticle coated orthodontic molar tubes (experimental) (Experimental): The nine orthodontic patients will receive 36 orthodontic molar tubes coated with ZnO nanoparticle in split-mouth cross quadrant manner, In each patient, two diagonal quadrants (i.e., upper right and lower left, or vice versa) will randomly assigned to each coated OMT and UOMT groups. evaluation will be after 2 weeks for microbial assessment biofilm in addition to plaque & gingival index. patients will be follow up for 3 month to evaluation bond failure rate.
  Interventions: Device: Zinc oxide nanoparticle coated orthodontic molar tubes (experimental)
- orthodontic molar tubes (control) (Placebo Comparator): The nine orthodontic patients will receive 36 the non-coated orthodontic molar tube in split-mouth cross quadrant manner, In each patient, two diagonal quadrants (i.e., upper right and lower left, or vice versa) will randomly assigned to each coated OMT and UOMT groups. evaluation will be after 2 weeks for microbial assessment biofilm in addition to plaque & gingival index. patients will be follow up for 3 month to evaluation bond failure rate.
  Interventions: Device: orthodontic molar tubes (control)

INTERVENTIONS:
Device: Zinc oxide nanoparticle coated orthodontic molar tubes (experimental) — nine orthodontic patients each one will receive 2 coated zinc oxide nanoparticle molar tubes in split-mouth manner and will assess for antimicrobial effect on s. mutans & lactobacillus after two weeks, in addition to evaluation of bond failure rate after three months.
  Arms: Zinc oxide nanoparticle coated orthodontic molar tubes (experimental)
Device: orthodontic molar tubes (control) — nine orthodontic patients each one will receive two uncoated molar tubes in split-mouth manner and will assess for antimicrobial effect on S. mutans & lactobacillus after two weeks, also, evaluation of the bond failure rate after three months period.
  Arms: orthodontic molar tubes (control)

SUMMARY:
Orthodontic treatment is an elective procedure to improve the patient's dentofacial appearance. The complex design of fixed appliances provides a platform that leads to increased plaque accumulation around orthodontic brackets. So, the risk to develop demineralization area adjacent to orthodontic brackets is a major barrier in achieving this goal. Oral hygiene is greatly complicated following the placement of fixed orthodontic Appliances. Molar tube in place are considered for nearly all patients experiencing fixed orthodontic therapy over the whole treatment period, which normally lasts 1.5 to 2 years. To the best of the authors' knowledge, the application and antimicrobial efficacy of zinc oxide (ZnO) nanoparticles coating on orthodontic molar tube material has not been integrated clinically. White spot lesions during orthodontic treatment have a documented etiology. Briefly, the accumulation of plaque and food around brackets, bands, wires, and other attachments caused decreased pH and increased S. mutans colonization, which led to the possibility of clinical demineralization.

The aims of study are to assess the antimicrobial effect of nanoparticle coated stainless steel orthodontic molar tube material (OMT) with zinc oxide (ZnO) nanoparticles in relative to uncoated orthodontic molar tube (UOMT) against the streptococcus. mutans& lactobacllius bacteria that cause white spot lesion around the fixed orthodontic appliance. .

DETAILED DESCRIPTION:
Aim:

The aim of this prospective randomized clinical trial is to assess the antimicrobial efficacy of nanoparticle coating stainless steel orthodontic molar tube (OMT) with zinc oxide (ZnO) nanoparticles in relative to uncoated orthodontic molar tube (UOMT).

Objectives:

1. Compare the antimicrobial properties of the zno nanoparticle coated OMT in relative to uncoated orthodontic molar tube (UOMT).
2. Evaluate and compare the clinical bond failure rate between the coated OMT and the UOMT. The null hypothesis is that there is no significant difference in the antimicrobial effects and the rate of bond failure between the non-coated and coated stainless steel orthodontic molar tube using ZnO NPs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are seeking or under orthodontic treatment with fixed appliances Subjects must be healthy &well fit medically.

  * Subjects with no signs or symptoms of oral mucosal disease.
  * Subjects should not receive oral antimicrobials or antibiotic therapy for more than 3 months prior to sample enrolling.
  * non-pregnant or lactating Female patient.
  * Subjects is not smokers

Exclusion Criteria:

* Patients with a greater tendency to accumulate plaque (e.g., having congenital anomalies such as cleft lip and palate) or undergo orthognathic surgery

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the antimicrobial Effect of ZnO Nanoparticles Coated orthodontic molar tube in relative to the uncoated orthodontic molar tube | After 2 weeks
  Compare the antimicrobial properties of the zno nanoparticle coated OMT in relative to uncoated orthodontic molar tube (UOMT), through taking swaps from patient and sent to laboratory to culturing swaps samples to evaluating the colony forming unit number of S. mutans&lactobacillus bacteria which consider mean cause of white spot lesion and compare with the uncoated orthodontic molar tube swaps cultures.

SECONDARY OUTCOMES:
Evaluate and compare the clinical bond failure rate between the coated orthodontic molar tube and the uncoated orthodontic molar tube | 3 months
  By following up patients for 3 months recording the bond failure occurs through out the this period with date and location of debond tubes for coated and uncoated orthodontic molar tubes.

CONTACTS AND LOCATIONS:
Overall Officials: Dhiaa Hu Al-Groosh, P.H.D, Study Director — University of Baghdad
Locations (1):
- University of Baghdad /college of dentistry, Baghdad, Bab Al Muadam, Iraq

IPD SHARING:
Plan to Share IPD: No
It will be mostly available on request.

REFERENCES:
- [Background] Cerroni S, Pasquantonio G, Condo R, Cerroni L. Orthodontic Fixed Appliance and Periodontal Status: An Updated Systematic Review. Open Dent J. 2018 Sep 28;12:614-622. doi: 10.2174/1745017901814010614. eCollection 2018. PMID 30369970
- [Background] Antonio-Zancajo L, Montero J, Albaladejo A, Oteo-Calatayud MD, Alvarado-Lorenzo A. Pain and Oral-Health-Related Quality of Life in Orthodontic Patients During Initial Therapy with Conventional, Low-Friction, and Lingual Brackets and Aligners (Invisalign): A Prospective Clinical Study. J Clin Med. 2020 Jul 3;9(7):2088. doi: 10.3390/jcm9072088. PMID 32635196
- [Background] Erbe C, Hornikel S, Schmidtmann I, Wehrbein H. Quantity and distribution of plaque in orthodontic patients treated with molar bands. J Orofac Orthop. 2011 Mar;72(1):13-20. doi: 10.1007/s00056-010-0001-4. Epub 2011 Mar 11. English, German. PMID 21484542
- [Background] Srivastava K, Tikku T, Khanna R, Sachan K. Risk factors and management of white spot lesions in orthodontics. J Orthod Sci. 2013 Apr;2(2):43-9. doi: 10.4103/2278-0203.115081. PMID 24987641
- [Background] Beyth N, Houri-Haddad Y, Baraness-Hadar L, Yudovin-Farber I, Domb AJ, Weiss EI. Surface antimicrobial activity and biocompatibility of incorporated polyethylenimine nanoparticles. Biomaterials. 2008 Nov;29(31):4157-63. doi: 10.1016/j.biomaterials.2008.07.003. Epub 2008 Aug 3. PMID 18678404
- [Background] Lim BS, Lee SJ, Lee JW, Ahn SJ. Quantitative analysis of adhesion of cariogenic streptococci to orthodontic raw materials. Am J Orthod Dentofacial Orthop. 2008 Jun;133(6):882-8. doi: 10.1016/j.ajodo.2006.07.027. PMID 18538253
- [Background] Shah AG, Shetty PC, Ramachandra CS, Bhat NS, Laxmikanth SM. In vitro assessment of photocatalytic titanium oxide surface modified stainless steel orthodontic brackets for antiadherent and antibacterial properties against Lactobacillus acidophilus. Angle Orthod. 2011 Nov;81(6):1028-35. doi: 10.2319/021111-101.1. PMID 22007663
- [Background] Abdulhussein, D. A. (2022). AN ANTIMICROBIAL NANOPARTICLES COATED FIXED ORTHODONTIC RETAINER (AN IN VITRO STUDY). University of Baghdad.